CLINICAL TRIAL: NCT04381273
Title: Oral Health and Psychosocial Factors During the Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Antonio Ciardo, Dr. med. dent., Heidelberg University
Other Study IDs: S-303/2020
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Covid-19; Periodontal Diseases; COVID
MeSH Terms: conditions — COVID-19; Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — questionnaire-based assessment

SUMMARY:
This prospective observational study examines the effects of the Covid-19 pandemic on oral health, taking psychosocial factors into account, and the possible impact of a high periodontitis risk on the severity of the need for treatment in Covid-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Residence in Germany
* Understanding of study participation and consent

Exclusion Criteria:

* <18 years old
* Residence outside of Germany

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The largest possible number of people should be given the opportunity to participate in this questionnaire considered the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1178 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
How do people assess their oral health-related quality of life in times of the Covid-19 pandemic? | 08.05.2020-31.07.2020
  The survey consists of validated and unvalidated items giving the opportunity to assess periodontitis risk, psychosocial stress, anxiety, depression and oral health related quality of life as well as questions focusing on experiences of the covid-19 pandemic.
Does the periodontitis risk have an influence on the severety of the Covid-19 disease and its' treatment? | 08.05.2020-31.07.2020
  The survey consists of validated and unvalidated items giving the opportunity to assess periodontitis risk, psychosocial stress, anxiety, depression and oral health related quality of life as well as questions focusing on experiences of the covid-19 pandemic.

SECONDARY OUTCOMES:
Do psychosocial stress factors in times of the Covid-19 pandemic have an impact on their oral health related quality of life? | 08.05.2020-31.07.2020
  The survey consists of validated and unvalidated items giving the opportunity to assess periodontitis risk, psychosocial stress, anxiety, depression and oral health related quality of life as well as questions focusing on experiences of the covid-19 pandemic.
Have people changed their oral hygiene practices in times of the Covid-19 pandemic? | 08.05.2020-31.07.2020
  The survey consists of validated and unvalidated items giving the opportunity to assess periodontitis risk, psychosocial stress, anxiety, depression and oral health related quality of life as well as questions focusing on experiences of the covid-19 pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ciardo, Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided